CLINICAL TRIAL: NCT04265300
Title: Nutrition, Urinary Markers and Sleep Habits in Children
Brief Title: Hydration Intervention in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Douglas J Casa, Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H19-212
Record Dates: First submitted 2020-02-03; First posted 2020-02-11 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Dehydration in Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention provided
- Creative Roots (Experimental): The intervention group will receive Creative Roots beverages and be instructed to have at least one drink (251mL) available at each meal (i.e. breakfast, lunch, and dinner) and drink as much as they would like throughout the day (i.e. ad libitum) of either Creative Roots or any other beverage they would normally consume. Subjects will be asked the keep their empty Creative Roots bottles to return them to the lab. Subjects will be instructed to refrigerate the beverages for better taste, and to refrigerate the beverages after opening.
  Interventions: Dietary Supplement: Creative Roots

INTERVENTIONS:
Dietary Supplement: Creative Roots — The Creative Roots beverage is a coconut water-based drink with three flavors Mixed Berry, Watermelon Lemonade, and Peach Mango. The ingredients are as follows and are the same for all three flavors: water, coconut water concentrate, citric acid, stevia leaf extract, natural flavor, rosemary extract (to preserve flavor). Contains: coconut
  Arms: Creative Roots

SUMMARY:
The investigators are conducting this research study to determine learn how daily habits and fluid choices impact children's health, sleep, cognitive function and mood. The investigators look to determine if a hydration intervention using an alternative beverage may impact these variables in children.

Maintaining an appropriate level of hydration throughout the day has multiple health benefits. Maintaining a desirable hydration status improves overall health and wellbeing (mood, reaction time, sleep quality, cognitive function, etc.) in adults, but negative health and mental effects of hypohydration are not fully understood in an adolescent population. Maintaining appropriate hydration in adolescents presents unique challenges with respect to schedule (e.g. the availability of fluid during the school day and after school activities) as well as ensuring the most beneficial beverage choice. Adolescents can be very meticulous regarding their preferred beverage (e.g. choosing a sugary drink over water) and parents prefer their children consume the healthiest option for their food and beverages, often times leading to conflict.

Therefore the purpose/goal of the proposed study is to determine if a hydration intervention using an alternative sweetened beverage will improve hydration and other overall health (e.g. cognitive function, sleep quality, mood etc.)

The investigators hypothesize, that by giving children an alternative tasty option, they will consume more fluids which may lead to improving and maintaining their chronic hydration state. Implementing a beverage intervention with a sweet alternative option (i.e. Creative Roots) could improve hydration levels in adolescents. In turn, possibly improving mood, reaction time, sleep quality, and cognitive function. All of which are vital in the overall development of the adolescent.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* aged 7-12 years old
* Guardians must also meet the criteria which is that

  * 1) they shop at Whole Foods, Costco, or Trader Joe's
  * 2) they use organic ingredients &
  * 3) they check the nutritional content on foods for their children.

Exclusion Criteria:

* prior diagnosis of cognitive or learning disabilities
* history of chronic kidney disease,
* diabetes
* sleep disorders
* use of medications that may alter water balance (e.g. diuretics, laxatives, antacids, anti-histamines, NSAIDs, blood pressure medication)
* mood and anxiety medications (e.g. antidepressants, anxiolytics, beta-blockers, ADHD medications).
* Other medications that can cause urine color changes include isoniazid, sulfasalazine, metronidazole, nitrofurantoin, amitriptyline, cimetidine, indomethacin, zaleplon, methocarbamol, metoclopramide, warfarin, rifampin, and phenazopyridine
* Participants who do not like the Creative Roots beverage

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Hydration Status Change | 7 weeks
  Change in WUT Score (Weight Urine and Thirst)

SECONDARY OUTCOMES:
Sleep Change | 7 weeks
  Change in quantity
Cognitive functioning Change | 7 weeks
  Change in Go-no-go test score
Cognitive functioning Change | 7 weeks
  Change in modified flanker task score
Mood Change | 7 weeks
  Change in Modified Mood Questionnaire Score

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No